CLINICAL TRIAL: NCT06288191
Title: A Phase 2, Open Label, Single Arm, Clinical Trial of Neoadjuvant Nivolumab and Relatlimab in Stage II To IV (M0) Resectable Cutaneous Squamous Cell Carcinoma
Brief Title: Neoadjuvant Nivolumab and Relatlimab in Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIA2023/490; CA224-1065 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2024-02-04; First posted 2024-03-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: neoadjuvant; immunotherapy; pathological response
MeSH Terms: interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Intervention Model Description: Open label, single arm, single centre, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): Nivolumab and relatlimab will be administered in a fixed dose combination (FDC). The dose and dosing regimen for this study is nivolumab 480 mg and relatlimab 160 mg - 2 vials per infusion. All patients are scheduled to receive two doses of nivolumab and relatlimab FDC prior to surgery on days 1 and 29. Patients without a complete pathological response to neoadjuvant therapy may receive standard of care radiotherapy per multidisciplinary team meeting discussion.
  Interventions: Drug: Nivolumab 240 mg / Relatlimab 80 mg in a fixed dose combination

INTERVENTIONS:
Drug: Nivolumab 240 mg / Relatlimab 80 mg in a fixed dose combination — Dual inhibition of the distinct LAG3 and PD-1 checkpoint pathways
  Other Names: Opdualag

SUMMARY:
The goal of this study is to test neoadjuvant therapy with the dual inhibition of Programmed cell death protein 1 (PD-1) and lymphocyte activation gene 3 (LAG-3) immune checkpoint pathways in a cohort of treatment-naïve, resectable stage II to IV cutaneous squamous cell carcinoma on the pathological response rate (pCR) and recurrence-free survival.

DETAILED DESCRIPTION:
This is a phase 2, open label, single cohort, single centre, clinical trial of neoadjuvant immunotherapy with dual inhibition of PD-1 and LAG-3 immune checkpoint pathways. The hypothesis is that neoadjuvant therapy produces a higher pathological response rate (pCR) and a longer recurrence-free survival in a cohort of treatment-naïve patients with resectable stage II to IV (M0) cutaneous squamous cell carcinoma compared to neoadjuvant cemiplimab monotherapy in Checkmate 358 (n=123, NCT02488759, historical control).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Written informed consent
3. Histologically confirmed, resectable stage II to IV cutaneous squamous cell carcinoma defined as:

   Non-head and neck cuSCC:
   1. stage II (T2, N0, M0)
   2. stage III (T3, N0, M0; or T1-3, N1, M0)
   3. stage IV (T1-3, N2 or N3, M0; or T4a or T4b, any N, M0)

   Cutaneous head and neck CC:
   1. stage II (T2, N0, M0)
   2. stage III (T3, N0, M0)
   3. stage IV (T4a or T4b, any N, M0)
4. In-transit metastases (ITM) are permitted if they are completely resectable. ITM defined as skin or subcutaneous metastases that are > 20 mm from the primary lesion but not beyond the regional nodal basin.
5. Measurable disease according to RECIST version 1.1 criteria (≥10 mm longest diameter for primary lesions and / or ≥10 mm in shortest diameter for lymph nodes as determined by CT imaging) within 2 weeks of the start of study treatment.
6. Tumour amenable to a newly obtained core biopsy of a lesion which has not been previously irradiated. Archival tissue from a past primary or nodal cuSCC lesion (if applicable) or tissue taken for current diagnosis will also be collected.
7. Previous radiotherapy permitted if performed at a prior site of disease not seen at baseline.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
9. Documented adequate haematological, hepatic, renal, and thyroid function determined by blood pathology
10. Anticipated life expectancy of > 12 months
11. Women of childbearing potential must have a negative serum pregnancy test within 24 hours of the first dose of study treatment or within 72 hours if this is not feasible. Effective contraception should be used for the duration of study treatment and for 5 half-lives (or 5 months) after the last dose. Egg donation (ova, oocytes) should be avoided for the same period. There are no partner-pregnancy or sperm donation avoidance requirements for male patients.

Exclusion Criteria:

1. Clinical or radiographic evidence of distant metastasis
2. SCC of the eyelid, vulva, penis and perianus
3. Any contraindication to the administration of nivolumab and / or relatlimab
4. Prior anti-PD-1, CTLA-4 (Cytotoxic T-lymphocyte associated protein 4), PDL-1 (Programmed death-ligand 1) or LAG 3 (Lymphocyte-Activation Gene 3) antibody exposure, or an agent directed to another stimulatory or co-inhibitory T-cell receptor for any disease or any chemotherapy or experimental local or systemic drug treatment
5. Active autoimmune disease or a requirement for chronic steroid therapy other than hormone replacement therapy

   The following are permitted:
   * Vitiligo
   * Type I diabetes mellitus on stable insulin therapy
   * Residual autoimmune hypothyroidism on stable hormone replacement
   * Resolved childhood asthma or atopy
   * Psoriasis not requiring systemic treatment
   * Autoimmune conditions which are not expected to recur in the absence of an external trigger.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment.

   The following are permitted:
   * Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.)
   * Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if patient is on a stable dose
   * Non-absorbed intra-articular steroid injections.
7. Known additional malignancies (unless adequately treated) active within the previous 3 years, except for locally curable cancers that have been apparently cured.

   The following malignancies, if undergone successful definitive resection or curative treatment, are permitted:
   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ, but excluding carcinoma in situ of the bladder) that have undergone potentially curative therapy
   * Prostatic intraepithelial neoplasia
   * In situ melanoma
   * Atypical melanocytic hyperplasia
   * Multiple primary melanomas
   * Other malignancies for which the patient has been disease free for 3 years, not requiring active anti-cancer therapy.
8. Uncontrolled or significant cardiovascular disease including, but not limited to any of the following:

   * Myocardial infarction (MI) or stroke/transient ischemic attack within the 6 months prior to consent
   * Uncontrolled angina within the 3 months prior to consent
   * Any history of clinically significant arrhythmias (such as poorly controlled atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
   * QTc (corrected QT interval) prolongation > 480 ms
   * History of other clinically significant cardiovascular disease (i.e. cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled venous thrombosis, etc)
   * Cardiovascular disease-related requirement for daily supplemental oxygen
   * History of 2 or more M.I.s OR 2 or more coronary revascularisation procedures (regardless of the number of stent placements during each procedure)
   * Patients with history of myocarditis, regardless of aetiology.
9. Troponin T (TnT) or I (TnI) >2 × institutional ULN (upper limit of normal). Participants with TnT or TnI levels between >1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤1 ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are <2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enrol the participant following cardiologist recommendation must be made to the Lead Investigator.
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis or current interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Has had an allogenic tissue/solid organ transplant
13. Has a known history of Human Immunodeficiency Virus (HIV). Note: no testing for HIV is required unless mandated by local health authority.
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
15. Pregnant or breast-feeding females
16. Concurrent medical or social conditions that may prevent the patient from attending assessments per schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | Week 6
  Proportion of patients with a pathological complete response, as determined on the week 6 surgical specimen using the guidelines published by the International Neoadjuvant Melanoma Consortium: Complete pathological response (pCR) = 0% viable tumour cells in the surgical specimen

SECONDARY OUTCOMES:
Pathological near pathological response (near pCR), partial response (pPR) and pathological non-response (pNR) rate | Week 6
  Proportion of patients with each non-pCR response category, as determined on the week 6 surgical specimen using the guidelines published by the International Neoadjuvant Melanoma Consortium (INMC):
  * Major pathological response (pCR + near-pCR),
  * Near complete pathological response - (near pCR) - >0% - ≤10% viable tumour
  * Partial pathological response (pPR) - >10 - ≤50% viable tumour
  * Non pathological response (pNR) - >50% viable tumour
Toxicity and tolerability of neoadjuvant immunotherapy and surgery | Week 24
  The proportion of patients with adverse events (AE) per Common Terminology Criteria for Adverse Events (CTCAE), from initiation of study treatment until at least 135 days after the end of treatment. Outcome measures include the proportion of patients with each of the following measures:
  1. An AE by CTCAE term / grade
  2. AEs attributable to neoadjuvant treatment
  3. Grade 3/4/5 AEs by AE term
  4. The duration of events reported in (a)
  5. Delayed study treatment and/or delay surgery due to an AE
  6. A requirement to discontinue study treatment early due to an AE
  7. Oral or parenteral steroid treatment for immune-related adverse events.
  8. Post-operative complications (e.g. seroma formation, wound infection or lymphoedema) and duration of events.
  9. Post-operative complications at 3 weeks and one year using the Clavien-Dindo Classification.
  10. Surgeon's assessment of 'operability' and morbidity from baseline and at surgery per INMC questionnaires.
Objective response rate to neoadjuvant therapy | Week 6
  The proportion of patients within each response category, as assessed using RECIST version 1.1, comparing week 6 to baseline CT and MRI.
  Objective response rate= CR and PR
Metabolic response rate to neoadjuvant immunotherapy | Week 6
  The proportion of patients within each response category, as assessed using the Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) and the standardised uptake value (SUV) comparing week 6 to baseline positron emission tomography (PET) scan.
  Metabolic response rate = Complete metabolic response (CMR) and partial metabolic response (PMR).
Recurrence-free survival | 10 years
  The proportion of patients alive and disease free from the time of surgery
Disease progression rate | Week 6
  The proportion of patients alive and with RECIST-defined progression of disease from the date of consent to the first radiographical evidence of local, regional or distant progression.
  Disease progression which leads to unresectable cutaneous squamous cell carcinoma (cuSCC)
Event-free survival rate | 10 years
  Proportion of patients with EFS defined as the earliest of any of the following events:
  1. Time from 1st dose study treatment to disease progression (unresectable stage III or stage IV disease),
  2. Time of surgery to recurrence of cuSCC (local, regional or distant)
  3. Treatment related death
  4. Disease related death
Overall survival | 10 years
  The proportion of patients alive at years 1, 2, 5 and 10, and to actual date of death (in months), from the first dose of study treatment.
Patient reported quality of life (QLQ-C30) | 1 year
  The published scoring for: The European Organization for the Research and Treatment of Cancer Quality of Life of Cancer Patients Questionnaire (QLQ-C30). A 30 item instrument where a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
  Changes in patient rated quality of life (QOL) scores using QLQ-C30 are recorded at baseline (within 7 days of first dose of study treatment) and at 6 -12 weekly intervals until the end of year 1 will be measured.
  The correlation of the QLQ-C30 scores with adverse events will be measured.
Patient reported quality of life (EQ-5L-5D) | 1 year
  The published scoring for: The European Quality of Life (EQ-5L-5D).
  Each dimension has 5 levels: no problems, some problems, extreme problems.
  The EQ visual analogue scale (VAS records) the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable, health state' and 'Worst imaginable health state'.
  Changes in patient rated quality of life (EQ-5D-5L) scores recorded at baseline (within 7 days of first dose of study treatment) and at 6 -12 weekly intervals until the end of year 1 will be measured.
  The correlation of the EQ-5L-5D scores with adverse events will be measured.
Study treatment completion rate and the causes of any missed treatments | Week 8
  Proportion of patients receiving full neoadjuvant drug treatment per schedule and number of treatments missed.
  Proportion of patients undergoing planned surgery at week 6. Reasons for incomplete study treatment e.g. adverse event, withdrawn consent, disease progression, patient lost to follow-up.
De-escalation of adjuvant radiotherapy. | Week 8
  Proportion of patients where adjuvant radiotherapy was planned at baseline but who did not need radiotherapy as a result of pathological response and pathologically clear surgical margins.

OTHER OUTCOMES:
Identification of tissue and blood biomarkers of response / resistance | 1 year
  Identification of biomarkers in tumour tissue and blood that may be predicitve of the response or resistance to neoadjuvant immunotherapy.
Profile of the gut microbiome from faecal samples and relationship to response and toxicities. | Week 6
  Identification of the type and abundance of gut microbes and the correlation with treatment response and incidence of treatment-related toxicities.
The pathological response to RECIST, immune related response criteria and PERCIST response | Week 6
  Proportion of patients with concordance across all tumour evaluations
Assessment of the response to neoadjuvant using the immune-related response criteria (irRC) and correlate the assessment with the RECIST 1.1 response at each timepoint | Week 6
  Bi-dimensional measurements of all target lesions per irRC guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Ines Da Silva, Principal Investigator — Melanoma Instiute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No